CLINICAL TRIAL: NCT04673942
Title: An Adapted Phase 2a/2b, Study to Evaluate the Safety, Tolerability, and Efficacy of AdAPT-001 in Subjects With Refractory Solid Tumors
Brief Title: A Study of AdAPT-001 in Subjects With Sarcoma and Refractory Solid Tumors
Acronym: BETA-PRIME
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: EpicentRx, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BETA-PRIME
Record Dates: First submitted 2020-12-08; First posted 2020-12-17 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Solid Tumor, Adult; Cancer; Neoplasms; Sarcoma; Sarcoma,Soft Tissue; Chondrosarcoma
Keywords: oncolytic virus; immunotherapy; adenovirus; intratumoral injection; AdAPT-001; Sarcoma
MeSH Terms: conditions — Neoplasms; Sarcoma; Chondrosarcoma; Adenoviridae Infections | interventions — Immune Checkpoint Inhibitors

STUDY DESIGN:
Intervention Model Description: The study is an exploratory open label single-arm interventional study using a 3 + 3 dose escalation safety run-in (PART 1) followed by a dose expansion single-agent (PART 2), followed by expansion (PART 3) single agent or single agent plus checkpoint inhibitor, followed by an adaptive designed Phase 2..
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- PART 1: Dose Escalation Safety Run-In (Enrollment Completed) (Experimental): Subjects will be treated with AdAPT-001 as a single injection, one time.
  Interventions: Biological: AdAPT-001
- PART 2: Dose Expansion Single-Agent (Enrollment Completed) (Experimental): 6 subjects will be enrolled in the Lead In Cohort. A Safety Analysis will be performed after 6 subjects have received at least 24 doses. Upon Safety team review as a continuous reassessment of safety, an additional 19 subjects may be enrolled. All subjects in PART 2 will receive injections of AdAPT-001 on Days 1 and 15 of 28-day cycles.
  Interventions: Biological: AdAPT-001
- PART 3: Expansion (Enrollment Completed) (Experimental): Up to 45 subjects will be enrolled in the expansion cohort to receive either AdAPT-001 on Days 1 and 15 of 28-day cycles or AdAPT-001 on Days 1 and 15 plus a checkpoint inhibitor of 28-day cycles.
  Interventions: Biological: AdAPT-001; Drug: Checkpoint Inhibitor, Immune
- Phase 2 (Enrollment Open) (Experimental): Approximately 55 to 80 subjects with advanced solid tumors including sarcoma to receive either AdAPT-001 on Days 1 and 15 of 28-day cycles or AdAPT-001 on Days 1 and 15 plus a checkpoint inhibitor of 28-day cycles..
  Interventions: Biological: AdAPT-001; Drug: Checkpoint Inhibitor, Immune

INTERVENTIONS:
Biological: AdAPT-001 — Oncolytic virus administered by intratumoral injection
Drug: Checkpoint Inhibitor, Immune — Checkpoint Inhibitor per investigator discretion based on diagnosis and subject tolerability
  Arms: PART 3: Expansion (Enrollment Completed); Phase 2 (Enrollment Open)

SUMMARY:
AdAPT-001 is an oncolytic virus that is injected directly into the tumor or via intraarterial administration. The purpose of this study is to find out if AdAPT-001 is safe and tolerable. The next step is to find out if AdAPT-001 if efficacious with or without a checkpoint inhibitor.

DETAILED DESCRIPTION:
This is a dose escalation protocol to determine, first and foremost, the safety, tolerability and feasibility of intratumoral administration of AdAPT-001.

The study has 3 parts. Different groups of patients will participate in each part.

PHASE 1 PART 1: Dose Escalation Safety Run-In (CLOSED - Enrollment Completed) During PART 1, all participants will be treated with AdAPT-001 as a single injection, one time. Participants will be assigned to different dose levels to find the highest dose of AdAPT-001 that is safe and tolerable.

PHASE 1 PART 2: Dose Expansion Single-Agent (CLOSED - Enrollment Completed) All participants in PART 2 will receive injections of AdAPT-001 on Days 1 and 15 of 28-day cycles.

PHASE 1 PART 3: Expansion (CLOSED - Enrollment Completed) Subjects will be assigned to the following two arms. If a checkpoint inhibitor is indicated for the subject, the subject may be enrolled on Arm 2 per investigator discretion, otherwise subjects may be enrolled on Arm 1.

Arm 1: Intratumoral administration of AdAPT-001 (1.0 x 10¹² viral particles) on Day 1 and 15 of each 28-day cycle for up to 12 injections.

Arm 2: Intratumoral administration of AdAPT-001 (1.0 x 10¹² viral particles) on Day 1 and 15 of each 28-day cycle for up to 12 injections plus a checkpoint inhibitor per investigator discretion

PHASE 2: (OPEN to Enrollment)

Subjects with advanced solid tumors will participate in a basket two-arm parallel group evaluation (Phase 2) where eligible participants will be assigned to the following two arms based on confirmed histology by the treating investigator.

Arm 1: Confirmed Histological Diagnosis of Sarcoma Intratumoral Administration of AdAPT-001 (1.0 x 10¹² viral particles) on Day 1 and 15 of each 28-day cycle for up to 12 injections with or without a checkpoint inhibitor.

Arm 2: Confirmed Histological Diagnosis of Advanced Solid Tumor indicated to receive at least one checkpoint inhibitor.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is capable of understanding the purpose and risks of the study and has provided written Informed Consent.
2. Subject is male or female, aged at least 18 years.
3. Subject has a histologically or cytologically confirmed diagnosis of an advanced malignant solid tumor(s) who have received all conventional therapies considered appropriate by Investigator and have a tumor that is easily accessible and/or palpable for treatment. Ultrasound guidance may be used to aid administration.
4. Subject's Eastern Cooperative Group (ECOG) performance status is 0-1 at Screening.
5. Subject has acceptable liver function at Screening, as evidenced by:

   1. Bilirubin < 1.5 x ULN (upper limit of normal)
   2. AST (SGOT) and ALT (SGPT) < 3.0 x ULN (upper limit of normal)
   3. Alkaline Phosphatase < 2.5 x ULN (upper limit of normal)
6. Subject has a Serum Creatinine < 1.5 x ULN (upper limit of normal)
7. Subject has acceptable hematologic status at Screening, as evidenced by:

   1. Absolute neutrophil count > 1,500 cells/mm3; > 1.5 x 109/L, and
   2. Platelet count > 75,000/mm3; > 75.0 x 109/L, and
   3. Hemoglobin (HGB) ≥ 8.0 g/dL; ≥ 5.6 mmol/L
8. Subject has an INR < 1.5
9. Female subjects of childbearing potential (i.e., women who have not been surgically sterilized or have not been post-menopausal for at least one year), and male subjects with partners of childbearing potential, must agree to use medically acceptable methods of contraception beginning on Study Day 1 and continuing until at least four weeks after administration of the subject's final dose of AdAPT-001. Medically acceptable contraception is defined as either: 1) usage by at least one of the partners of a barrier method of contraception, together with usage by the female partner, commencing at least three months prior to Study Day 1, of a stable regimen of any form of hormonal contraception or an intra-uterine device, or 2) usage by the couple of a double-barrier method of contraception. Use of a single-barrier method alone or abstinence alone is not considered adequate.
10. Subject is willing and able to comply with all protocol procedures, evaluations and rescue measures.
11. OPTIONAL: Archival formalin-fixed paraffin-embedded block(s) or previously cut archival tissue for at least 5 unstained slides (if available).

Exclusion Criteria:

1. Presence of a serious co-morbid medical condition, or a clinically significant laboratory finding(s) that, in the opinion of the Investigator, suggests the presence of an infectious, endocrine, and/or other inadequately treated systemic disorder.
2. A known uncontrolled active bacterial, fungal, or viral infection. No subject with an active SARS-CoV-2 infection (within 14 days of a positive test)
3. Known positive history of human immunodeficiency virus (HIV) test
4. Subjects who have active hepatitis.
5. If female, subject is pregnant and/or breastfeeding.
6. Subjects with active autoimmune disease or history of autoimmune disease that might recur and may affect vital organ function or require immune suppressive treatment including systemic corticosteroids, should be excluded.

   Note: Subjects in any condition requiring systemic treatment with corticosteroids (prednisone > 10 mg/day or equivalent of the similar drug) or other immunosuppressive agents within 14 days before AdAPT-001), but currently or previously treated with any of the following steroid regimens were included: Topical, ophthalmic, intra-articular, intranasal, or inhaled corticosteroids with minimal systemic absorption; prophylactic short-term use of corticosteroids.
7. Prior adenoviral therapy for any indication except vaccination against infectious disease. Subjects receiving COVID-19 or live vaccination, cannot start treatment until 7 days after completing the vaccination. Recommend waiting at least 28 days from AdAPT-001 dose prior to receiving COVID-19 vaccination. Concurrent treatment with Evusheld is allowed.
8. Chemotherapy or immunotherapy within 14 days of study treatment. Hormonal therapy (including tamoxifen, aromatase inhibitors, and gonadotropin releasing hormone agonists) is allowed. Concurrent treatment with bisphosphonate and RANK ligand inhibitor is allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2021-03-29 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicities (DLT) | 28 days
  All subjects in PART 1 will be assessed for the development of dose-limiting toxicity (DLT) during treatment with AdAPT-001. The DLT assessment period is defined as: Day of Injection through 28 days post injection (Safety Follow Up). A DLT will be defined as any Grade 3 or higher adverse event, as assessed by the National Cancer Institute Common Toxicity Criteria for Adverse Events (CTCAE) version 5.0.
Maximum tolerated dose | 28 days
  In PART 1, A MTD is determined if any cohort experiences 2 subjects with DLT's.
Safety of a multiple dose regimen of AdAPT-001 | 6 months
  The safety data will include adverse events, serious adverse events, performance status, clinical laboratory tests, vital signs and physical examination results.
Anti-tumor activity of the two-arm dose regimens of AdAPT-001 in Phase 2 | 6 months
  To evaluate the efficacy of the two-arm dose regimens of AdAPT-001 in subjects with advanced solid tumors that have progressed after treatment with standard therapies or for which there are no appropriate therapies available as measured by durable (≥4 months) stable disease per Response Evaluation Criteria in Solid Tumors (RECIST).

SECONDARY OUTCOMES:
Anti-tumor activity of AdAPT-001 | 6 months
  In PART 2 and PART 3, overall response rate (ORR) and best overall response rates per response evaluation criteria outlined in Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1), as well as progression-free survival (PFS), and duration of response will be assessed.
Objective response rate | 6 months
  Preliminarily to assess anti-tumor activity of AdAPT-001 by objective response rates (ORR) and best overall response rates per response evaluation criteria outlined in RECIST guideline (Version 1.1),

OTHER OUTCOMES:
Anti-tumor activity by iRECIST | 6 months
  ORR and best overall response rates per Immune Response Evaluation Criteria in Solid Tumors (iRECIST)
Biodistribution | 6 months
  This outcome will measure TGFβ trap concentrations in the serum and, in patients who consent to tissue collections, test for TGFβ trap expression in the treated tumors.

CONTACTS AND LOCATIONS:
Overall Officials: Bryan Oronsky, MD PhD, Study Director — EpicentRx, Inc.
Locations (6):
- United States (6):
  - City of Hope, Duarte, California
  - California Cancer Associates for Research and Excellence, cCARE, San Marcos, California
  - Providence Saint John's Health Center, Santa Monica, California
  - Cleveland Clinic, Cleveland, Ohio
  - Mary Crowley Cancer Research, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Derived] Reid TR, Oronsky B, Williams J, Caroen S, Conley A. TGF-beta trap of AdAPT-001 turns up the heat on tumors and turns down checkpoint blocker resistance. J Immunother Cancer. 2024 Oct 26;12(10):e009613. doi: 10.1136/jitc-2024-009613. PMID 39461878
- [Derived] Kesari S, Bessudo A, Gastman BR, Conley AP, Villaflor VM, Nabell LM, Madere D, Chacon E, Spencer C, Li L, Larson C, Reid T, Caroen S, Oronsky B, Stirn M, Williams J, Barve MA. BETA PRIME: Phase I study of AdAPT-001 as monotherapy and combined with a checkpoint inhibitor in superficially accessible, treatment-refractory solid tumors. Future Oncol. 2022 Sep;18(29):3245-3254. doi: 10.2217/fon-2022-0481. Epub 2022 Aug 11. PMID 35950603